CLINICAL TRIAL: NCT02314663
Title: Effectiveness of a Combined Strategy to Improve Therapeutic Compliance and Degree of Control Among Patients With Hypercholesterolaemia: a Randomised Clinical Trial
Brief Title: Effectiveness of a Combined Strategy to Improve Therapeutic Compliance and Degree of Control Among Patients With Hypercholesterolaemia
Acronym: EFESCOM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Gerencia de Atención Primaria, Albacete (Other)
Collaborators: Instituto de Salud Carlos III (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GAPALBACETE
Record Dates: First submitted 2014-12-04; First posted 2014-12-11 (Estimated); Last update posted 2014-12-11 (Estimated); Status verified 2014-12

CONDITIONS: Hypercholesterolemia; Medication Adherence; Primary Health Care
Keywords: hypercholesterolaemia; medication adherence; primary health care
MeSH Terms: conditions — Hypercholesterolemia; Medication Adherence

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention group (Experimental): "COMBINED STRATEGY" (a + b + c). Participants in the intervention group will be supplied with: a) "printed matter"; b) "mobile-telephone text messages"; and, c) "self-report cards".
  This group receive routine recommendations from their GPs, in accordance with current European clinical practice guidelines on the management of hypercholesterolaemia and cardiovascular risk
  Interventions: Device: "COMBINED STRATEGY"
- Control group (No Intervention): This group receive routine recommendations from their GPs, in accordance with current European clinical practice guidelines on the management of hypercholesterolaemia and cardiovascular risk

INTERVENTIONS:
Device: "COMBINED STRATEGY" — Participants in the intervention group will be supplied with: a) "printed matter" containing information on the disease and its management (this will be handed out at each of the follow-up visits); b) "mobile-telephone text messages" containing guideline summaries, reminders of forthcoming appointments and/or arrangements for making new appointments in the event of non-attendance (in the periods between visits); and, c) "self-report cards" to check compliance with recommendations (across the entire follow-up).
  Arms: Intervention group

SUMMARY:
Background In subjects with hypercholesterolaemia, cholesterol values remain above guideline levels. One of the limiting factors to the achievement of goals in such patients is therapeutic non-adherence. The aim of this study is to assess the effectiveness of an intervention designed to improve control of hypercholesterolaemic patients, consisting of a combined strategy that would include the delivery of printed information, treatment-compliance check cards and the dispatch of text messages as complementary measures in support of the intervention at the general practitioner's practice.

Methods/Design A randomised, parallel-group clinical trial will be conducted at the family medicine outpatient facilities of eight health centres in three of Spain's Autonomous Regions, covering a total of 358 subjects aged 18 years or over with diagnosis of hypercholesterolaemia. Patients in the intervention group will be supplied with printed material with information on the disease and its management, mobile-telephone text messages with guideline summaries, reminders of forthcoming appointments and/or arrangements for making new appointments in the event of non-attendance, and self-report cards to check compliance with recommendations. Both groups -intervention and control- will receive routine recommendations from their physicians in accordance with current European clinical practice guidelines for hypercholesterolaemia and cardiovascular risk management. As regards the measurements to be made, the main variable is the proportion of subjects who attain the low density lipoprotein cholesterol levels set as a target across a follow-up period of 24 months. The secondary variables are as follows: adherence to recommendations on lifestyle and adherence to drug treatment; variation in lipid profiles and cardiovascular risk levels; appearance of cardiovascular events; physical activity; food consumption; smoking habit; anthropometric measures; blood pressure; health problems; use of hypolipidaemic agents; socio-demographic data; beliefs and expectations about preventive recommendations; and degree of satisfaction with the combined strategy.

Discussion Should this intervention prove effective, a recommendation could be issued on the application of this combined strategy to subjects with hypercholesterolaemia. It is a simple, relatively inexpensive intervention.

ELIGIBILITY:
Inclusion Criteria:

* be diagnosed with hypercholesterolaemia, as defined according to the criteria stipulated in the cardiovascular prevention guidelines of the 2009 Prevention Activities and Promotion of Health Programme (total cholesterol of 250 mg/dl or higher).
* be patients aged 18 years or over attending any of the participating health centres.

Exclusion Criteria:

* any person hindered from participating in the follow-up of the proposed intervention, e.g., illiterate subjects and non-users of mobile telephones.
* any person with a physical disability or impairment which prevents him/her from attending the follow-up visits.
* any person suffering from a significant chronic organic or psychiatric disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 358 (Estimated)
Dates: Start 2013-01; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
The proportion of subjects who attain the LDL-C levels set as targets by the Guidelines for Management of Dyslipidaemias and CVR | 24 months
  The main study variable is the proportion of subjects who attain the LDL-C levels set as targets by the Guidelines for Management of Dyslipidaemias and CVR, across a follow-up period of 24 months. The plasma values taken as cardiovascular prevention targets are: a) LDL-C <100 mg/dl for patients without established cardiovascular disease or diabetes mellitus; and, b) LDL-C <70 mg/dl for patients with diabetes mellitus or established cardiovascular disease

SECONDARY OUTCOMES:
adherence to lifestyle guidelines and adherence to drug treatment | 24 months
  adherence to lifestyle guidelines and adherence to drug treatment, as seen from self-reported adherence (adapted Haynes-Sackett test), validated questionnaire (Morisky-Green test) and Likert scale with 5 response options
variation in plasma lipid profile levels | 24 months
  variation in plasma lipid profile levels (total cholesterol, LDL-C, HDL-C and triglycerides
variation in cardiovascular risk level | 24 months
  SCORE and REGICOR tables will be used for the evaluation
Occurrence of cardiovascular events | 24 months
  Ischaemic heart disease, atherothrombotic cerebrovascular disease, heart failure and peripheral artery disease
determination of the frequency of food consumption | 24 months
  determination of the frequency of food consumption
smoking habit (answers affirmatively to the question, "Do you smoke?") | 24 months
  smoking habit, with a smoker being defined as anyone who answers affirmatively to the question, "Do you smoke?"
physical activity (degree of aerobic physical exercise performed (active, partially active or inactive) | 24 months
  physical activity, i.e., determination of the degree of aerobic physical exercise performed (active, partially active or inactive)
anthropometric measures (i.e., weight, height, body mass index (BMI), and waist circumference) | 24 months
  i.e., weight, height, body mass index (BMI), and waist circumference
systolic and diastolic blood pressure | 24 months
  systolic and diastolic blood pressure (two measurements), with the result being the mean of the two results
degree of satisfaction with the combined strategy ((Likert scale with 5 response options ranging from 1 "very dissatisfied" to 5 "very satisfied") | 24 months
  degree of satisfaction with the combined strategy according to a satisfaction questionnaire (Likert scale with 5 response options ranging from 1 "very dissatisfied" to 5 "very satisfied").
health problems (WONCA ICPC-2 classification) | 24 months
  health problems
use of hypolipidaemic drug treatment | 24 months
  use of hypolipidaemic drug treatment (type of drug and dose)

CONTACTS AND LOCATIONS:
Overall Officials: Ignacio Párraga-Martínez, PhD, Principal Investigator — Health Care Service of Castilla-La Mancha

REFERENCES:
- [Background] European Association for Cardiovascular Prevention & Rehabilitation; Reiner Z, Catapano AL, De Backer G, Graham I, Taskinen MR, Wiklund O, Agewall S, Alegria E, Chapman MJ, Durrington P, Erdine S, Halcox J, Hobbs R, Kjekshus J, Filardi PP, Riccardi G, Storey RF, Wood D; ESC Committee for Practice Guidelines (CPG) 2008-2010 and 2010-2012 Committees. ESC/EAS Guidelines for the management of dyslipidaemias: the Task Force for the management of dyslipidaemias of the European Society of Cardiology (ESC) and the European Atherosclerosis Society (EAS). Eur Heart J. 2011 Jul;32(14):1769-818. doi: 10.1093/eurheartj/ehr158. Epub 2011 Jun 28. PMID 21712404
- [Background] Kotseva K, Wood D, De Backer G, De Bacquer D, Pyorala K, Keil U; EUROASPIRE Study Group. Cardiovascular prevention guidelines in daily practice: a comparison of EUROASPIRE I, II, and III surveys in eight European countries. Lancet. 2009 Mar 14;373(9667):929-40. doi: 10.1016/S0140-6736(09)60330-5. PMID 19286092
- [Background] Vegazo O, Banegas JR, Civeira F, Serrano Aisa PL, Jimenez FJ, Luengo E; Estudio HISPALIPID. [Prevalence of dyslipidemia in outpatients of the Spanish health service: the HISPALIPID Study]. Med Clin (Barc). 2006 Sep 9;127(9):331-4. doi: 10.1157/13092314. Spanish. PMID 16987452
- [Background] Marrugat J, Solanas P, D'Agostino R, Sullivan L, Ordovas J, Cordon F, Ramos R, Sala J, Masia R, Rohlfs I, Elosua R, Kannel WB. [Coronary risk estimation in Spain using a calibrated Framingham function]. Rev Esp Cardiol. 2003 Mar;56(3):253-61. doi: 10.1016/s0300-8932(03)76861-4. Spanish. PMID 12622955
- [Background] Perk J, De Backer G, Gohlke H, Graham I, Reiner Z, Verschuren M, Albus C, Benlian P, Boysen G, Cifkova R, Deaton C, Ebrahim S, Fisher M, Germano G, Hobbs R, Hoes A, Karadeniz S, Mezzani A, Prescott E, Ryden L, Scherer M, Syvanne M, Scholte op Reimer WJ, Vrints C, Wood D, Zamorano JL, Zannad F; European Association for Cardiovascular Prevention & Rehabilitation (EACPR); ESC Committee for Practice Guidelines (CPG). European Guidelines on cardiovascular disease prevention in clinical practice (version 2012). The Fifth Joint Task Force of the European Society of Cardiology and Other Societies on Cardiovascular Disease Prevention in Clinical Practice (constituted by representatives of nine societies and by invited experts). Eur Heart J. 2012 Jul;33(13):1635-701. doi: 10.1093/eurheartj/ehs092. Epub 2012 May 3. No abstract available. PMID 22555213
- [Background] Kotseva K, Wood D, De Backer G, De Bacquer D, Pyorala K, Keil U; EUROASPIRE Study Group. EUROASPIRE III: a survey on the lifestyle, risk factors and use of cardioprotective drug therapies in coronary patients from 22 European countries. Eur J Cardiovasc Prev Rehabil. 2009 Apr;16(2):121-37. doi: 10.1097/HJR.0b013e3283294b1d. PMID 19287307
- [Background] Waters DD, Brotons C, Chiang CW, Ferrieres J, Foody J, Jukema JW, Santos RD, Verdejo J, Messig M, McPherson R, Seung KB, Tarasenko L; Lipid Treatment Assessment Project 2 Investigators. Lipid treatment assessment project 2: a multinational survey to evaluate the proportion of patients achieving low-density lipoprotein cholesterol goals. Circulation. 2009 Jul 7;120(1):28-34. doi: 10.1161/CIRCULATIONAHA.108.838466. Epub 2009 Jun 22. PMID 19546386
- [Background] Bermingham M, Hayden J, Dawkins I, Miwa S, Gibson D, McDonald K, Ledwidge M. Prospective analysis of LDL-C goal achievement and self-reported medication adherence among statin users in primary care. Clin Ther. 2011 Sep;33(9):1180-9. doi: 10.1016/j.clinthera.2011.07.007. Epub 2011 Aug 12. PMID 21840055
- [Background] De Geest S, Sabate E. Adherence to long-term therapies: evidence for action. Eur J Cardiovasc Nurs. 2003 Dec;2(4):323. doi: 10.1016/S1474-5151(03)00091-4. No abstract available. PMID 14667488
- [Background] Banegas JR, Lopez-Garcia E, Dallongeville J, Guallar E, Halcox JP, Borghi C, Masso-Gonzalez EL, Jimenez FJ, Perk J, Steg PG, De Backer G, Rodriguez-Artalejo F. Achievement of treatment goals for primary prevention of cardiovascular disease in clinical practice across Europe: the EURIKA study. Eur Heart J. 2011 Sep;32(17):2143-52. doi: 10.1093/eurheartj/ehr080. Epub 2011 Apr 6. PMID 21471134
- [Background] Marquez Contreras E, Casado Martinez JJ, Corchado Albalat Y, Chaves Gonzalez R, Grandio A, Losada Velasco C, Obando J, de Eugenio JM, Barrera JM. [Efficacy of an intervention to improve treatment compliance in hyperlipidemias]. Aten Primaria. 2004 May 15;33(8):443-50. doi: 10.1016/s0212-6567(04)79430-5. Spanish. PMID 15151791
- [Background] McDonald HP, Garg AX, Haynes RB. Interventions to enhance patient adherence to medication prescriptions: scientific review. JAMA. 2002 Dec 11;288(22):2868-79. doi: 10.1001/jama.288.22.2868. PMID 12472329
- [Background] Haynes RB, McKibbon KA, Kanani R, Brouwers C, Oliver T: Interventions to assist patients to follow prescriptions for medications. In: Cochrane Collaboration: Cochrane Library. Oxford: Update Software, 1998.
- [Derived] Parraga-Martinez I, Rabanales-Sotos J, Lago-Deibe F, Tellez-Lapeira JM, Escobar-Rabadan F, Villena-Ferrer A, Blasco-Valle M, Ferreras-Amez JM, Morena-Rayo S, del Campo-del Campo JM, Ayuso-Raya MC, Perez-Pascual JJ. Effectiveness of a combined strategy to improve therapeutic compliance and degree of control among patients with hypercholesterolaemia: a randomised clinical trial. BMC Cardiovasc Disord. 2015 Jan 19;15:8. doi: 10.1186/1471-2261-15-8. PMID 25599690